CLINICAL TRIAL: NCT05986422
Title: Phase 2a, Double-blind, Randomized, Placebo-controlled Trial of Methylprednisolone Versus Placebo in Patients with Cognitive Deficits in Post-COVID-19 Syndrome (PCS)
Brief Title: Methylprednisolone in Patients with Cognitive Deficits in Post-COVID-19 Syndrome (PCS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Heinrich J Audebert, Deputy Director of the Department of Neurology with Experimental Neurology at Charite Campus Benjamin Franklin, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PoCoVIT; 01EP2201 (Other Grant/Funding Number: BMBF)
Record Dates: First submitted 2023-08-09; First posted 2023-08-14 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-02

CONDITIONS: Post-COVID-19 Syndrome
Keywords: Long COVID; Cognitive deficits
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Cognition Disorders | interventions — Methylprednisolone

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-Blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylprednisolone (Active Comparator): Tested IMP: Methylprednisolone (film-coated tablet). Authorization status: Not authorized in this targeted therapeutic indication; methylprednisolone is authorized for treatment of multiple autoimmune diseases. The tablets being administered in this trial are an official trade product provided by the marketing authorization holder JenaPharm.
  Administration: Tablet containing 16 mg/tablet will be administered orally and according to bodyweight groups. Treatment period comprises 6 weeks of blinded daily IMP (investigational medicinal product) intake (verum or placebo) and 6 weeks of unblinded daily intake of Methylprednisolone. The general IMP titration regimen was investigated and proven to be safe in patients with cerebral vasculitis (Schirmer et al., 2020).
  Interventions: Drug: Methylprednisolone
- Placebo (Placebo Comparator): Comparator IMP: Placebo (film-coated tablet). Authorization status: Not authorized. To ensure identical conditions with the verum (Methylprednisolone), we will use placebo tablets of the same color and size in identical tablet packages for both the verum and placebo.
  Administration: Tablets (7 mm) will be administered orally and according to bodyweight groups. To achieve consistent conditions with the verum, titration will be conducted in a manner similar to the tested IMP (Methylprednisolone). Treatment period comprises 6 weeks of blinded daily IMP intake (placebo or verum) and 6 weeks of unblinded daily intake of Methylprednisolone.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — The treatment period consists of six weeks of daily intake of either Methylprednisolone or placebo (depending on randomization), followed by an additional six weeks of daily intake of open-label Methylprednisolone. During the study, follow-up assessments will be conducted at two points: at week 8 and week 20 from the start of each treatment phase.

SUMMARY:
This clinical trial aims to learn about the therapeutic value of Methylprednisolone, a well-known immunosuppressant, on cognitive deficits in patients with post-COVID-19 syndrome (PCS). The main questions it aims to answer are: 1) Does Methylprednisolone improve memory function in PCS patients compared to placebo? 2) Does Methylprednisolone improve other patient centered outcomes in PCS patients such as fatigue, mood and quality of life compared to placebo? 3)What are the side effects of Methylprednisolone in this patient population, and how common are they? Participants in this study will be patients with PCS and cognitive deficits, who will be asked to participate for 52 weeks. They will be randomly assigned to one of two groups: One group will receive Methylprednisolone once daily for six weeks, with a dosage reduction after week 4. The other group will receive a matching placebo once daily for six weeks, following the same titration regimen to ensure blinding. Participants will attend outpatient follow-up visits in weeks 8 and 20, with a final telephone follow-up after 52 weeks. Clinical examinations and safety monitoring will be conducted during the treatment phase. This study's results may help develop more effective therapies for this condition.

DETAILED DESCRIPTION:
Around 10-40% of mild COVID-19 patients experience persisting or new symptoms known as post-COVID-19 syndrome (PCS). Neurological symptoms, particularly cognitive deficits and fatigue, are common in PCS, with a higher prevalence in female patients (Boesl et al., 2021; Ceban et al., 2022). The underlying causes of PCS remain unclear, but some evidence suggests autoimmune mechanisms may play a role. Currently, there are no proven treatments for PCS, leading to a need for effective therapies. This randomized controlled trial (RCT) aims to investigate the impact of methylprednisolone, a generally well-tolerated and affordable drug, on cognitive deficits in PCS patients with suspected autoimmune involvement.

The objective is to demonstrate improvement in memory satisfaction as measured by the Multifactorial Memory Questionnaire (MMQ) in patients with post-COVID-19 syndrome treated with Methylprednisolone compared with placebo. Methylprednisolone is a well-known immunosuppressant used for multiple diseases of (suspected) autoimmune etiology.

This is a two-arm, double-blind, randomized, placebo-controlled trial evaluating the effects of Methylprednisolone versus placebo in patients with post-COVID-19 syndrome (PCS) and cognitive deficits. The study spans 52 weeks, and participants will be stratified based on age, sex, and cognitive screening using the Montreal Cognitive Assessment Scale (MoCA). They will be randomly assigned in a 1:1 ratio to receive either Methylprednisolone (including a tapering phase) or placebo for 6 weeks, followed by an additional 6 weeks of open treatment phase with Methylprednisolone after a 6-weeks treatment pause. During the study, follow-up visits will be conducted as outpatient visits in weeks 8 and 20, with a final telephone follow-up after 52 weeks. The screening and baseline examinations will involve recording of medical history, checking inclusion and exclusion criteria, and conducting clinical examinations. The intervention group will receive approximately 1mg/kg body weight oral Methylprednisolone once daily for 6 weeks, with dosage reduction after week 4. The other group will receive a matching placebo once daily for 6 weeks, following the same titration regimen to maintain blinding. The starting dose for both interventions will be Methylprednisolone at approximately 1 mg/kg body weight or matching placebo once per day. Throughout the treatment phase, all participants will undergo safety and monitoring examinations.

This clinical trial is of significant importance as it has the potential to benefit individuals with post-COVID-19 syndrome (PCS) by exploring the effects of Methylprednisolone on cognitive impairment and fatigue. Additionally, it may provide crucial insights into PCS's pathophysiological processes, leading to the development of more effective therapies and improved patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* History of confirmed (PCR or serology) SARS-CoV-2 infection according to WHO criteria
* Ongoing symptoms of PCS for ≥ 3 months
* Self-reported cognitive deficits at screening
* Male or female adult who is 18 years or older at the time of informed consent
* Subject is willing, understanding and able to provide informed consent
* Signed informed consent prior to initiation of any trial related measure
* For female subject or divers subjects:

  1. Confirmed post-menopausal state, defined as amenorrhea for at least 12 months, or
  2. If being of childbearing potential:

     1. Negative highly sensitive urine or serum pregnancy test before inclusion, and
     2. Practicing a highly effective birth control method (failure rate of less than 1%)

Exclusion Criteria:

* Any ongoing central nervous system disease
* Any major psychiatric disease within the last 10 years
* Previous medical history of gastric ulcer, osteoporosis and/or previous vertebral fractures, rheumatological disease or metabolic disease including diabetes mellitus
* Ongoing immunosuppressive therapy
* Patient is pregnant or breastfeeding at screening
* MMQ memory satisfaction subdomain >50 points at Screening
* Current malignant disease (including space-occupying brain tumors)
* Body weight <45kg
* Severe lactose intolerance
* Participation in another clinical interventional trial within the last 3 months or five half- lives of the other trial's IMP, if longer than 6 months previous to informed consent
* Patient is institutionalized by order of court or public authority
* Patient who might be dependent on the sponsor, the investigator or the trial site
* Place of living does not allow the subject to attend the planned study visits
* Other conditions that are likely to affect to safety of the study treatment (e.g., severely impaired immune status)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in memory satisfaction as measured by the Multifactorial Memory Questionnaire (MMQ) | 8 weeks after first IMP intake
  The MMQ is a participant-reported measure of memory satisfaction. It consists of three scales measuring separate aspects of metamemory including memory satisfaction, memory ability, and memory strategy. For memory satisfaction, eighteen items are rated on a 5-point Likert scale based on the test taker's experience over the previous two weeks.The score range is 0 to 72, with higher scores indicating a higher degree of satisfaction. A change of 13 points is commonly rated as clinically significant change. In this study, intra-patient change in MMQ subdomain memory satisfaction by ≥15 points from baseline to week 8 will be interpreted as meaningful improvement.

SECONDARY OUTCOMES:
Long-term improvement in memory satisfaction as measured by the Multifactorial Memory Questionnaire (MMQ) | 20 and 52 weeks after first IMP intake
  Intra-patient change in MMQ subdomain memory satisfaction from baseline to week 20, from week 8 to week 20 and from week 20 to week 52 will be documented.
Improvement in memory ability and memory strategy as measured by the Multifactorial Memory Questionnaire | 8 and 20 weeks after first IMP intake
  As secondary outcomes the MMQ subdomains memory ability and memory strategy are assessed. The memory ability subscale evaluates participants' self-perception of everyday memory capabilities. Participants are asked to rate the frequency with which they experience 20 common memory mistakes over the preceding two weeks. Scores on this subscale range from 0 to 80, where higher scores indicate better self-reported memory ability. The memory strategy subscale evaluates the usage of practical memory strategies and aids in day-to-day life. Respondents rate the frequency of their utilization of 19 memory strategies during the past two weeks. Scores on this subscale range from 0 to 76, with higher scores reflecting a greater implementation of memory strategies. Mean difference in MMQ subdomain 'memory ability' and 'memory strategy' from baseline to week 8 and to week 20 and from week 8 to week 20 will be documented.
Improvement in neurocognitive functions as measured by the Montreal Cognitive Assessment (MoCA) | 8 and 20 weeks after first IMP intake
  The MoCA is a sensitive and validated cognitive screening tool to test subjects quickly and accurately for mild cognitive impairment, irrespective of etiology. A person can gain a maximum of 30 points, and professionals consider a score of 26 or above to be normal. A score of 25 points or less may indicate some degree of cognitive impairment (18-25 = mild cognitive impairment, 10-17 = moderate cognitive impairment, fewer than 10 points = severe cognitive impairment). Intra-patient change in neurocognitive functions from baseline to week 8 and to week 20 and from week 8 to week 20 will be documented.
Improvement in neurocognitive functions as measured by the symbol digit modalities test (SDMT) | 8 and 20 weeks after first IMP intake
  The SDMT (oral version) detects cognitive impairment in less than five minutes and will be used to assess change in cognitive function over time. SDMT is a validated and established measure of cognition in multiple sclerosis capturing impairments such as processing speed and working memory, visual search and scanning, and oculomotor functioning. Patients are provided a sheet with nine symbols, each paired with a number on top of the page. The remainder of the page consists of a randomized, sequential assortment of these symbols. Participants are asked to respond verbally with the number corresponding to each symbol. The final score is the correct number of substitutions in 90s (range 0 to 110, higher score = higher neurocognitive function). Intra-patient change in neurocognitive functions from baseline to week 8 and to week 20 and from week 8 to week 20 will be documented.
Improvement in quality of life (QoL) as measured by the PROMIS questionnaire | 8, 20, and 52 weeks after first IMP intake
  The PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS measures can be used with the general population and with individuals living with chronic conditions. Intra-patient change in PROMIS score from baseline to week 8, week 20, and week 52 and from week 8 to week 20 will be documented.
Improvement in physical and mental fatigue as measured by the Chalder Fatigue Scale | 8, 20, and 52 weeks after first IMP intake
  The Chalder Fatigue Scale measures the extent and severity of tiredness and has been used in multiple randomized trials of behavioral interventions in patients with ME/CFS. Each of the 11 items is answered on a 4-point scale with an overall score ranging from 0 (asymptomatic) to 33 (maximum symptomology). Intra-patient change in physical and mental fatigue from baseline to week 8, week 20, and week 52 and from week 8 to week 20 will be documented.
Improvement in fatigue as measured by the Fatigue Severity Score (FSS) | 8, 20, and 52 weeks after first IMP intake
  The FSS is a 9-item scale that measures the severity of fatigue and its effect on a person's activities and lifestyle. Answers are scored on a seven-point scale (1 = strongly disagree; 7 = strongly agree). Thus, the minimum score is 9 (no fatigue), and the highest is 63 (heavy fatigue). Intra-patient change in fatigue severity from baseline to week 8, week 20, and week 52 and from week 8 to week 20 will be documented.
Improvement in mood as measured by the Becks Depression Inventory (BDI-II) | 8, 20, and 52 weeks after first IMP intake
  The BDI-II is a widely used self-report questionnaire designed to assess the severity of depression symptoms in individuals aged 13 years and older. It consists of 21 multiple-choice items, each corresponding to a specific symptom of depression. Respondents rate the intensity of their symptoms on a scale ranging from 0 to 3, with higher scores indicating greater levels of depression. Intra-patient change in mood from baseline to week 8, week 20, and week 52 and from week 8 to week 20 will be documented.
Difference of occurring AE and SAE comparing Methyprednisolone with placebo (IMP safety). | 8 and 20 weeks after first IMP intake
  Occurrence of IMP side and adverse effects, including but not limited to infections, endocrinologic disorders, and psychiatric complications, assessed with AE, SAE and SUSAR reports.

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Audebert, Prof., MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schirmer JH, Aries PM, Balzer K, Berlit P, Bley TA, Buttgereit F, Czihal M, Dechant C, Dejaco C, Garske U, Henes J, Holle JU, Holl-Ulrich K, Lamprecht P, Nolle B, Moosig F, Rech J, Scheuermann K, Schmalzing M, Schmidt WA, Schneider M, Schulze-Koops H, Venhoff N, Villiger PM, Witte T, Zanker M, Hellmich B. [S2k guidelines: management of large-vessel vasculitis]. Z Rheumatol. 2020 Nov;79(Suppl 3):67-95. doi: 10.1007/s00393-020-00893-1. No abstract available. German. PMID 33156399
- [Background] Boesl F, Audebert H, Endres M, Pruss H, Franke C. A Neurological Outpatient Clinic for Patients With Post-COVID-19 Syndrome - A Report on the Clinical Presentations of the First 100 Patients. Front Neurol. 2021 Sep 16;12:738405. doi: 10.3389/fneur.2021.738405. eCollection 2021. PMID 34603189
- [Background] Ceban F, Ling S, Lui LMW, Lee Y, Gill H, Teopiz KM, Rodrigues NB, Subramaniapillai M, Di Vincenzo JD, Cao B, Lin K, Mansur RB, Ho RC, Rosenblat JD, Miskowiak KW, Vinberg M, Maletic V, McIntyre RS. Fatigue and cognitive impairment in Post-COVID-19 Syndrome: A systematic review and meta-analysis. Brain Behav Immun. 2022 Mar;101:93-135. doi: 10.1016/j.bbi.2021.12.020. Epub 2021 Dec 29. PMID 34973396